CLINICAL TRIAL: NCT00815425
Title: Consortium for the Longitudinal Evaluation of African-Americans With Early Rheumatoid Arthritis (CLEAR) Registry
Brief Title: Consortium for the Longitudinal Evaluation of African Americans With Early Rheumatoid Arthritis (The CLEAR Registry)
Acronym: CLEAR
Status: Completed | Type: Observational
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: N01 AR002278; N01AR62278-6-0-1 (NIH)
Record Dates: First submitted 2008-12-29; First posted 2008-12-30 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Rheumatoid Arthritis
Keywords: African American
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, including DNA and serum, and urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- African Americans with RA: 1063 participants with RA
- African-Americans without RA: 550 participants without RA

SUMMARY:
Rheumatoid arthritis (RA) is a long-term autoimmune disease that is characterized by pain, stiffness, inflammation, swelling, and sometimes destruction of joints. RA usually requires lifelong treatment, including medications, physical therapy, exercise, education, and possibly surgery, but the course and severity of the disease can differ significantly from person to person. The purpose of this study is to identify genetic and other factors that determine the severity of RA in African Americans.

DETAILED DESCRIPTION:
RA is a chronic condition that causes inflammation of the joints and surrounding tissues. Symptoms may include pain, stiffness, swelling, and sometimes destruction of joints. RA can affect any joint, but it is most common in the wrist and fingers. More women than men get RA, and it often starts between the ages of 25 and 55. The course and severity of the disease can differ significantly from person to person. Some people with RA may have the disease for only a short time, or their symptoms might come and go, but the severe form of RA can last a lifetime. The purpose of this study is to identify genetic and other factors that determine the severity of RA in African Americans.

Participants in this study will include African Americans with RA and healthy African Americans with RA. There are two arms: (1) longitudinal; and (2) cross-sectional. The longitudinal arm has completed enrollment and is still in the follow-up phase. This consists of visits at baseline (less than 2 years disease duration; 3 years disease duration; and 5 years disease duration).

For the cross-sectional arm, there will be one study visit for all participants, which will last approximately 1 to 2 hours for participants without RA (controls) and 2 to 3 hours for participants with RA. For all participants, this visit will include a medical history review; questionnaires regarding health, functional ability, family, education, and work history; and blood and urine collection. For participants with RA, this visit will also include examination of the joints for pain and swelling, X-rays of the hands and feet, and a physical examination.

The urine samples will be stored for future analyses of protein and chemical markers. The blood samples will be used in three different ways: (1) isolation of DNA; (2) isolation of serum and plasma; and (3) isolation of RNA. Part of the blood samples will be used by the investigators to identify genes or proteins that may predispose people to develop RA or that may influence disease outcome or treatment response. If participants agree, their blood cells will be put through a procedure called immortalization, which will provide researchers with sufficient DNA for all future studies associated with this study and for other related projects. If the immortalization process fails, participants may be asked for an additional blood sample with which to repeat the procedure. However, participants will not be provided with any information on their genes.

ELIGIBILITY:
Inclusion Criteria for Group 1 Participants:

* Rheumatoid arthritis
* Self-declared as African American

Exclusion Criteria for Group 1 Participants:

* Lupus

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: African Americans with and without RA
Sampling Method: Non-Probability Sample
Enrollment: 1613 (Actual)
Dates: Start 2000-09; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Radiographic severity of rheumatoid arthritis in African Americans | Measured at any point during the duration of disease

CONTACTS AND LOCATIONS:
Overall Officials: S. Louis Bridges, Jr, MD, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States